CLINICAL TRIAL: NCT01706445
Title: Combined Inspiratory Muscle and 'Whole Muscle' Training in Children With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Collaborators: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other)
Responsible Party: Principal Investigator, Alejandro Lucia, MD PhD, Universidad Europea de Madrid
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: kid'strainingCF; CFtraining (Registry Identifier: PS09/00194)
Record Dates: First submitted 2012-10-09; First posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; exercise; children; cardiorespiratory fitness; muscle strength; pulmonary function; quality of life
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention)
- intervention (Other): Exercise training
  Interventions: Other: Other

INTERVENTIONS:
Other: Other — inspiratory muscle training (IMT) + aerobic and strength training 8-week duration IMT twice a day (mostly at home) + 3 weekly sessions of inhospital resistance + aerobic training
  Other Names: Exercise training
  Arms: intervention

SUMMARY:
To study the effects of an 8-week combined inspiratory muscle training and exercise (resistance+aerobic) program on of a lung volume, inspiratory muscle strength (maximal inspiratory pressure, PImax) and cardiorespiratory fitness (maximal oxygen uptake, VO2peak) (primary outcomes)and dynamic muscle strength, body composition and quality of life (QoL) in children with Cystic Fibrosis (CF) (secondary outcomes).

DETAILED DESCRIPTION:
The investigators hypothesized that the combined training program would significantly benefit most of the aforementioned variables (especially, primary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* boy/girl aged 6-17 years
* living in the Madrid area

Exclusion Criteria:

* severe lung deterioration [forced expiratory volume (FEV1) <50% of expected]
* unstable clinical condition (hospitalization within the previous 3 months)
* Burkholderia cepacia infection
* any disorder (e.g. muscle-skeletal) impairing exercise.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
cardiorespiratory fitness (VO2peak) | this outcome will be assessed up to 12 weeks
  maximum oxygen uptake (VO2peak), which is the best indicator of aerobic fitness in humans and an independent mortality predictor in children with cystic fibrosis

SECONDARY OUTCOMES:
quality of life | this outcome will be assessed up to 12 weeks
  children's QoL with the Spanish Version (1.0) of the Cystic Fibrosis Questionnaire-Revised (CFQ-R).

OTHER OUTCOMES:
Maximal inspiratory pressure (PImax) | september 2011-july 2012
  an indicator of the strength of inspiratory muscles

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Infantil Universitario Niño Jesús, Madrid, Madrid, Spain